CLINICAL TRIAL: NCT07219979
Title: Evaluating the Effectiveness of Remote Monitoring for Post-Operative Management of Distal Radius Fractures: A Randomized Controlled Trial
Brief Title: Evaluating the Effectiveness of Remote Monitoring for Post-Operative Management of Distal Radius Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Daniel London, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2127568
Record Dates: First submitted 2025-10-20; First posted 2025-10-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Distal Radius Fracture; Distal Radius Fracture Fixation
Keywords: distal radius fracture; postoperative follow-up; remote monitoring; virtual care; orthopaedic surgery
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two distinct groups and each group receives its respective intervention throughout the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring Follow-Up (Experimental): Participants in this arm will complete postoperative follow-up through a digital health platform. At 6 weeks, 3 months, and 6 months after surgery, they will complete electronic PROMs , measure grip strength using a dynamometer, and submit short wrist range-of-motion videos for remote evaluation. Participants will be instructed to contact the clinical team if any concerns arise.
  Interventions: Behavioral: Remote Monitoring Follow-Up
- In-Person Standard Follow-Up (Active Comparator): Participants in this arm will attend routine postoperative clinic visits at 6 weeks, 3 months, and 6 months, following standard of care for distal radius fracture management. At each visit, PROMs will be completed, and grip strength and range of motion will be measured by the clinical team. Care decisions and management will follow institutional standards for in-person postoperative evaluation
  Interventions: Behavioral: Standard In-Person Follow-Up

INTERVENTIONS:
Behavioral: Remote Monitoring Follow-Up — Participants will complete postoperative assessments through a secure, HIPAA-compliant digital health platform.
  Arms: Remote Monitoring Follow-Up
Behavioral: Standard In-Person Follow-Up — Participants will attend routine in-person postoperative clinic visits.
  Arms: In-Person Standard Follow-Up

SUMMARY:
This randomized controlled trial evaluates whether remote monitoring can provide a safe and effective alternative to traditional in-person follow-up after surgical fixation of distal radius fractures. The study compares functional outcomes, patient satisfaction, and complication rates between patients who receive virtual follow-up care and those who attend standard in-person visits.

DETAILED DESCRIPTION:
This single-center, randomized controlled trial investigates the feasibility, safety, and effectiveness of a virtual postoperative follow-up model for patients undergoing operative fixation of distal radius fractures. Following surgery, eligible adult patients will be randomized 1:1 to either (1) standard in-person follow-up or (2) remote monitoring.

Participants in the remote arm will complete follow-up assessments through secure online surveys, including PROMIS Upper Extremity, PROMIS-29, APEX, and ICHOM questionnaires. Grip strength will be measured using a dynamometer, and wrist range of motion will be evaluated through patient-submitted videos analyzed by the research team. Patients in the in-person arm will undergo identical assessments during routine clinic visits.

The trial is designed as a non-inferiority study powered to determine whether remote follow-up achieves comparable recovery outcomes to in-person care while potentially improving access, satisfaction, and efficiency. Safety monitoring will include review of all adverse events and complications, with predefined criteria for pausing or modifying the protocol if unexpected risks arise

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* Operatively treated distal radius fracture
* Access to smartphone/computer.

Exclusion Criteria:

* Prior significant wrist/hand injury
* lack of internet access
* Surgeon determination that injury is not suitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Upper Extremity Score | Baseline and 6 months
  The PROMIS Upper Extremity (UE) Computer Adaptive Test assesses upper limb function, including strength, dexterity, and ability to perform daily activities. Scores range from 0 to 100, with higher scores indicating better function. The primary analysis will compare mean change in PROMIS UE scores from baseline (2 weeks post-operation) to 6 months post-operation

SECONDARY OUTCOMES:
PROMIS-29 Score | Baseline and 6 months
  The PROMIS-29 Profile assesses global physical, mental, and social health across domains including pain interference, fatigue, physical function, depression, anxiety, and sleep. Scores range from 0-100, with higher scores reflecting better health status for positively scored domains.
Ambulatory Patient Experience Score | Baseline and 6 months
  The Ambulatory Patient Experience (APEX) Questionnaire measures patient satisfaction and experience with outpatient care using validated multi-item scales. Scores are transformed to a 0-100 scale, with higher scores indicating greater satisfaction
Grip Strength | Baseline and 6 months
  Grip strength will be measured using a standardized, FDA-cleared hand dynamometer in kilograms
Wrist Range of Motion | Baseline to 6 months
  Wrist flexion, extension, pronation, and supination will be measured using standardized photogoniometry methods. For remote participants, motion will be assessed via patient-submitted videos analyzed by study staff.
Complication Rate | From enrollment to the end of treatment at 6 months
  Complications including infection, hardware failure, malunion, nonunion, and stiffness will be recorded for all participants through chart review and patient report. Rates will be compared between the remote monitoring and in-person groups to ensure patient safety and equivalence of outcomes. Complications will be measured as a percentage of patients who experience the complication

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. London, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This study involves clinical and patient-reported data collected within a single institution (University of Missouri) under IRB-approved protocols that limit data use to authorized study personnel. While aggregate results will be disseminated through peer-reviewed publications and presentations, individual-level data will not be shared externally to protect participant privacy and comply with institutional data governance policies